CLINICAL TRIAL: NCT01858298
Title: Conservative Versus Non-conservative Treatment for Severe Dental Caries in Preschool Children and Its Impact on Oral Health-related Quality of Life, Anthropometric Measures, Space Loss and Anxiety: a Randomized Clinical Trial
Brief Title: Conservative Versus Non-conservative Treatment for Severe Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University College, London (Other); Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Jenny Abanto, Post-doctoral student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: usp; 2013/10330-8 (Other Grant/Funding Number: Processo FAPESP)
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Dental Caries
Keywords: Dental caries; Quality of Life; Pulpectomy; Tooth extraction
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulpectomy (Experimental): The technique of pulpectomy will be performed in one appointment according to clinical guidelines and followed by a composite resin crown.
  Interventions: Other: Conservative treatment: pulpectomy and composite resin crown
- tooth extraction (Experimental): The technique of tooth extraction of primary teeth will be performed according to clinical guidelines
  Interventions: Other: Non-conservative treatment: Tooth extraction

INTERVENTIONS:
Other: Conservative treatment: pulpectomy and composite resin crown
  Arms: pulpectomy
Other: Non-conservative treatment: Tooth extraction
  Arms: tooth extraction

SUMMARY:
The purpose of this study is to compare the effectiveness of the conservative (pulpectomy) versus non-conservative treatment (tooth extraction) of primary molars affected with severe dental caries associated to oral health-related quality of life, anthropometric and clinical outcomes.

DETAILED DESCRIPTION:
Treatment: evaluate two interventions for treating severe dental caries in primary molared of preschool children.

SAMPLE: preschool children aged 3 to 5 years with severe dental caries (SDC) in primary molars. SDC will be indicated by the Pufa index. The Pufa index records the presence of severely decayed teeth with visible pulp involvement (p), ulceration of the oral mucosa owing to root fragments (u), fistula (f) and abscess (a). Children with pufa-score > 0 in primary molars will be included in the study. All children aged 3 to 5 years, who sought dental screening at the Dental School, University of São Paulo (USP) in August to October 2013 can be initially eligible.

CLINICAL GROUPS RANDOMLY ASSIGNED:

* Group A: Conservative treatment represented by pulpectomies + teeth restoration with composite resin crown.
* Group B: Dental extraction

  * Treatment of carious teeth with pufa score =0 will receive dental fillings (01 occlusal surface affected: ART; 02 surfaces affected: composite resin; ≥ 03 surfaces affected: composite resin crown).
  * One operator (specialists in paediatric dentistry) blinded to the outcomes will carry out the treatments.

FOLLOW-UP: 4, 8 and 12 months.

OUTCOMES: All outcomes will be assessed by a single person interviewer/examiner blinded to the oral treatments groups.

1. Oral Health-Related Quality of Life:

   * Brazilian SOHO-5
   * Brazilian ECOHIS
2. Anthropometric measures:

   * Weight-for-age Z-score (WAZ)
   * Height-for-age Z-score (HAZ)
   * BMI-for age Z-score (BAZ)
3. Dental anxiety (Facial Image Scale).
4. Dental pain (Wong-Baker Scale)
5. Problems in the developing occlusion: loss of space

ELIGIBILITY:
Inclusion Criteria:

* Preschool children with severe dental caries (SDC) in primary molars.
* SDC will be indicated by the Pufa index
* The Pufa index records the presence of severely decayed teeth with visible pulp involvement (p), ulceration of the oral mucosa owing to root fragments (u), fistula (f) and abscess (a). Children with a pufa-score > 0 will be included in the study.

Exclusion Criteria:

* Children with severe crowding of anterior teeth
* Severe arch length deficiencies
* Children with systemic and neurological diseases or those with illnesses that adversely affect growth according to parents reports
* Children on regular nutrition supplements
* Children who had undergone dental treatment in the last three months and who were not willing to participate in the study. Tooth with anomalies, extensive crown destruction and impossibility of absolute isolation in the conservative intervention group.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
oral health-related quality of life | 12 months
  - OHRQoL instruments: Brazilian SOHO-5 Brazilian ECOHIS

SECONDARY OUTCOMES:
anthropometric measures | 12 months
  * Weight-for-age Z-score (WAZ)
  * Height-for-age Z-score (HAZ)
  * BMI-for age Z-score (BAZ)
loss of space | 12 months
  Extraction space The referent space was determined by measuring the distance between the mesial and distal midpoints of the adjacents teeth to extraction or pulpectomy
dental anxiety | 12 months
  Scale anxiety using the Facial Image Scale
Dental pain | 12 months
  The Wong-Baker Faces Pain Scale will be used to asses dental pain

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Abanto, PhD, Principal Investigator — University of Sao Paulo